CLINICAL TRIAL: NCT05960500
Title: All on Six Versus Parallel Implant Distribution for Screw Retained Maxillary Fixed Single Denture Opposing Mandibular All on Four Implant Distribution
Brief Title: All on Six Versus Parallel Implant Distribution for Maxillary Denture Opposing Mandibular All on Four
Acronym: ASPISRMSDOMF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mennat Elrahman Essam Eldeen, Assistant Lecturer, Mansoura University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A05080622
Record Dates: First submitted 2023-06-18; First posted 2023-07-25 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Peri-Implantitis; Occlusal Trauma; Implant Complication
Keywords: soft tissue changes; occlusal stability; implant stability
MeSH Terms: conditions — Peri-Implantitis | interventions — Drug Implants

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Six implants in parallel distribution (Active Comparator): patients received 6 implants in parallel distribution in anterior, premolar and molar region
  Interventions: Procedure: implant
- Six implants according to all on six concept (Active Comparator): patients recived four axially placed anterior Implants(*General system) in lateral and first premolar region and two distally tilted 30 degree posteriorly in molar region relative to the occlusal plane supporting screw retained maxillary single denture.
  Interventions: Procedure: implant

INTERVENTIONS:
Procedure: implant — All on six versus parallel implant distribution
  Other Names: prothesis

SUMMARY:
Thirty maxillary edentulous patients with previous mandibular All-on-4 screw retained prosthesis and their age ranged from 55 to 65 years were selected from the outpatient clinic, of prosthodontics Department, Faculty of Dentistry, Mansoura University from March 2022 to July2022 and 80% power was used to calculate patients sample according to the results of a previous study 1 which showed no significant difference was reported when comparing occlusal stability ,implant stability and periimplant soft tissue changes between different implants angulation of both groups. (Effect size=.70mm and α=.05). The power analysis was performed using the G*Power program (version 3.1.5, Kiel, Germany)

DETAILED DESCRIPTION:
the aim of this study is to compare between All-on-Six distributed dental implants "Anterior 4 Implant Parallel and Posterior 2 Implant Distally Tilted" versus parallel distribution supporting screw retained maxillary single denture regarding soft tissue changes around implants, implant stability and occlusal stability.

The primary outcome is to study implant stability and occlusal stability. The secondary outcome is to evaluate periimplant soft tissue changes. The null hypothesis of this study will be there is no difference between the two studied groups.All patients were informed about the proposal of this study, the line of treatment, and the need for regular and frequent recalls. Their acceptance to participate in this study was confirmed and they signed the consent form of the ethical committee of the faculty of dentistry. This study gained the approval of the ethical committee of the Faculty of Dentistry, with approval number (A05080622).

all the patients were divided randomly into two equal groups as follows Group I patients received four axially placed anterior Implants(*General system) in lateral and first premolar region and two distally tilted 30 degree posteriorly in molar region relative to the occlusal plane supporting screw retained maxillary single denture.

Group II patients received 6 implants in parallel distribution in anterior, premolar and molar region

ELIGIBILITY:
Inclusion Criteria:

* patient with maxillary edentulous alveolar ridges.
* patient complained from insufficient retention and stability of their maxillary single denture.

Exclusion Criteria:

* medically compromised patients.
* patients with parafunctional habits.

Ages: 55 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-06-05 (Actual); Primary Completion 2023-05-10 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
soft tissue changes around implants | 1 year
  The distance between marginal gingiva and the tip of the probe was measured using a calibrated plastic periodontal probe this distance is considered as pocket depth (PD).Probing depth was evaluated at buccal, lingual, mesial and distal aspect of each implant. using a calibrated pressure sensitive plastic periodontal probe.

SECONDARY OUTCOMES:
occlusal stability | 1 year
  - Evaluation of the the concentration, changes of occlusion and visualization of the masticatory pressure conditions and amount of occlusal wear occured by Digital Occlusal Analyzer System (OccluSense)
implant stability | 1year
  - Evaluation of the rate of Implant stability A range of PTVs (- 6 to +2) was considered for integrated implants that was measured by periotest device*. The hand piece was. held perpendicular to the long axis of the implants.

CONTACTS AND LOCATIONS:
Overall Officials: Mennat Elrahman Essam Eldeen, Phd, Principal Investigator — Mansoura university Faculty of Dentistry Prosthodontics Department
Locations (1):
- Mansoura university, Al Mansurah, Dakahlya, Egypt

IPD SHARING:
Plan to Share IPD: No
. Evaluation was done for all patients at three evaluation periods as follows: T0: immediately before screwing the final prosthesis.T6: 6 months after unscrewing of the final prosthesis.T12: 12 months after unscrewing of the final prosthesis.